CLINICAL TRIAL: NCT02510781
Title: A Study on Neoadjuvant Therapy for Her-2 Positive Breast Cancer and the Prognosis Detecting Circulating Tumor Cells
Brief Title: A Study on Neoadjuvant Therapy for Her-2 Positive Breast Cancer and the Prognosis by Detecting CTCs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Affiliated to Military Medical Science, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJ307-Neo02
Record Dates: First submitted 2015-07-23; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Docetaxel; Trastuzumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A group (Experimental): docetaxel+carboplatin+trastuzumab
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Carboplatin
- B group (Active Comparator): Epirubicin+docetaxel+trastuzumab-docetaxel+trastuzumab
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Epirubicin — 75mg/m2 d1 evry 21days
  Other Names: pharmorubicin
  Arms: B group
Drug: Docetaxel — 75mg/m2 d1 evry 21days
  Other Names: Taxotere
Drug: Trastuzumab — 6mg/kg(loading dosage is 8mg/kg)
  Other Names: Herceptin
Drug: Carboplatin — Area Under Curve(AUC)=6 d1 evry 21days
  Other Names: Paraplatin
  Arms: A group

SUMMARY:
Docetaxel plus carboplatin and trastuzumab has been a standard treatment for patients with human epidermal growth factor receptor-2（HER-2）positive. The investigators witnessed a higher pathological complete remission(pCR) rate but no obvious increase in cardiac toxicity when used the anthracycline instead of carboplatin. The investigators expect to carry out a large sample size clinical research to optimize the existing therapeutic regimen

ELIGIBILITY:
Inclusion Criteria:

* 18≤aged<70
* pathologic diagnosis of invasive breast cancer，staging ii to iii，the diameters≥2cm indicated by MRI or axillary lymph node（+）
* Immunohistochemical（IHC） positive for 3+ or FISH（+）
* clear hormone receptor（HR） status
* Eastern cooperative oncology group(ECOG)=0/1
* LVEF≥55%
* pathologic grading of Miller and Payne
* screening laboratory values with the following parameters：absolute neutrophils acount：≥1500/mm3,total bilirubin:≤2.0×ULM,Aspartate transaminase (AST)/ALT≤2.5×ULM,platelet≥80000/mm3，serum creatinine≤1.5×ULM
* no pregnant or nursing
* signed Informed consent forms

Exclusion Criteria:

* prior exposure to any treatments for breast cancer
* inflammatory/Bilateral/IV stage breast cancer
* poor physical condition
* pregnant or nursing
* Cardiac risk（Congestive heart failure、arrhythmia、myocardial infarct、Refractory hypertension（systolic pressure>180mmHg/diastolic pressure>100mmHg））
* any other cancer within 5 years prior to screening with the exception of cervical carcinoma and non melanoma skin cancer
* Allergic to chemotherapy drugs

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | up to one year

SECONDARY OUTCOMES:
clinical response rate | up to one year
Number of Adverse Event | up to one year

CONTACTS AND LOCATIONS:
Overall Officials: zefei jiang, Ph.D, Principal Investigator — Academy MMS,China
Locations (1):
- Hospital affiliated to military medical science, Beijing, Beijing Municipality, China